CLINICAL TRIAL: NCT07139340
Title: Does the Use of HA Gel Following Third Molar Extraction Decrease the Incidence of Alveolar Osteitis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A300816
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2016-08

CONDITIONS: Alveolar Osteitis
MeSH Terms: conditions — Dry Socket

STUDY DESIGN:
Intervention Model Description: Control group (No HA gel), and study group (HA gel)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (HA gel) (Active Comparator): HA gel was placed intrasocket after extraction
  Interventions: Other: HA gel
- Control group (No HA gel) (No Intervention): Nothing was placed intrasocket after extraction

INTERVENTIONS:
Other: HA gel — Hyaluronic Acid gel 0.8% 1 mL
  Other Names: Hyaluronic Acid gel
  Arms: Study group (HA gel)

SUMMARY:
The study aimed to investigate the effectiveness of Hyaluronic Acid gel on decreasing the incidence of alveolar osteitis after mandibular third molar extraction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients (ASA=1)
* Patients need extraction of mandibular third molar
* Patients can attend recalls

Exclusion Criteria:

* Smoking patients
* Patients taking oral contraceptive pills
* Bad oral hygiene

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Occurence of Alveolar Osteitis (AO) | 7 postoperative days
  Presence of empty extraction socket without healing clot indicates AO (measured by clinical inspection; Presence of AO=1, Absence of AO=0)

SECONDARY OUTCOMES:
Postoperative pain | 7 postoperative days
  Presence of postoperative pain (measured by Visual Analogue Scale (VAS) from 0 (least pain) to 10 (worst pain))

CONTACTS AND LOCATIONS:
Locations (1):
- Delta university for science and technology, Gamasa, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No